CLINICAL TRIAL: NCT03266315
Title: Probiotics Supplementation and Intestinal Microbiome in Neonates With Gastrointestinal Surgery
Acronym: ProPS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Manufacturer discontinued the product used for the study: Business decision
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Belal Alshaikh, Clinical Associate Professor, Department of Pediatrics, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: REB16-2401
Record Dates: First submitted 2017-08-24; First posted 2017-08-30 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Probiotics; Infant, Newborn; Surgical Procedures, Operative; Gastro-Intestinal Disorder
MeSH Terms: conditions — Digestive System Diseases | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): subjects will be randomly assigned to receive FloraBaby
  Interventions: Biological: FloraBaby
- Placebo (Placebo Comparator): subjects will be randomly assigned to receive placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: FloraBaby — 1 sachet will be added to a minimum of 1 mL of brest milk, sterile water or formula (in formula fed babies) once a day
  Other Names: Probiotics
  Arms: Probiotics
Other: Placebo — 1 sachet will be added to a minimum of 1 mL of brest milk, sterile water or formula (in formula fed babies) once a day
  Arms: Placebo

SUMMARY:
Congenital defects of the gastrointestinal tract commonly require surgical intervention in the neonatal period. Intestinal surgery during this critical period of microbiome acquisition results in aberrant colonization of the gastrointestinal tract by several pathways. Surgical stress is known to cause disruption of the gut barrier and increase intestinal permeability and bacterial translocation. This process triggers exaggerated immune responses that lead to inflammation and sometimes infectious complications. Post-operative use of antibiotics has been shown to potentiate the growth of pathogenic bacterial species Adults with abdominal surgery who received post-op probiotics reported a significant reduction in surgical site infection, urinary tract infection, and combined infection. Currently, probiotics used only in the non-surgical population of infants.

The main objective of this study is to determine the impact of probiotics administration on the intestinal microbiome in neonates undergoing intestinal surgery.

DETAILED DESCRIPTION:
Research Objectives/Question:

The main objective of this study is to determine the impact of probiotics administration on the intestinal microbiome in neonates undergoing gastrointestinal surgery.

Primary question:

Diversity and abundance of stool microbiome at after 1 and 3 weeks of initiation of probiotics

Secondary outcomes:

1. Length of hospital stay

Methodology:

Study design This study will be a randomized controlled double-blinded trial in the NICU at Alberta Children's Hospital. Probiotics or placebo will be administered orally or via naso- or orogastric feeding tube. Intestinal microbiome data will be compared between the two groups. The study duration will be 24 months.

Study Population Infants born between 23 - 41 weeks of gestation, admitted to NICU at Alberta Children's Hospital for gastrointestinal surgery.

1. Inclusion Criteria:

   1. Infants born between 23 - 41 weeks of gestation
   2. Required gastrointestinal surgery in the first week of life (including spontaneous intestinal perforation, bowel atresia, mechanical bowel obstruction, volvulus, gastroschisis)
   3. Ready to start enteral feeding
2. Exclusion Criteria:

   1. Infants with major congenital anomalies excluding gastrointestinal tract 3. Palliative care patients 4. Septic babies with positive blood, CSF or urine culture

   Sample Size and feasibility:

   Connivant sample of 20 patients (10 in each group)

   Study protocol. Infants will be identified within 48 hours of surgery and parents will be approached for informed consent. Once consent is obtained, subjects will be randomly assigned to receive either probiotics or placebo. Investigators will conduct the randomization using a computer-generated table of random numbers generated at the University of Calgary.

   Preparation and Administration of Study Drug The study supplementation will be started at the when oral feeds will reach 24 mL/kg/day after surgery after collecting a stool/ostomy sample. The decision to start feeding will be made by the neonatal and surgical team. After the first stool/ostomy sample is obtained, one study sachet to a minimum of 1 mL of Expressed Breast Milk (EBM) (mothers own milk or donor human milk) once a day.

   Placebo sachet will be made of 0.3 g maltodextrin and be administered to the control group in the same manner. If the infant is placed NPO, the study drug will be stopped and restarted together with refeeding. Both probiotics and placebo will be packaged as a single-dose sachet. The study probiotic/placebo will be given till discharge. If the infant is transferred outside NICU, the study drug will be dispensed with the infant and clinical outcomes will be ascertained in collaboration with the local Pediatrician at the time of infants' discharge home.

   Sample collection Nurses will collect the stool samples at 3-time points: prior to initiation, 1 week after and 3 weeks after probiotic or placebo administration is commenced. "Stool" will be collected directly from the infant's ostomy bag and diaper with a sterile spatula. As soon as a sample is collected, the nurse will contact the investigators. The samples will then be placed in a laboratory freezer (-80°C) within 24 hours of collection. Batched samples will be transported to the University of Calgary Genomics laboratory for subsequent microbiome processing.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born between 23 - 41 weeks of gestation
2. Required gastrointestinal surgery (including spontaneous intestinal perforation, bowel atresia, mechanical bowel obstruction, volvulus, gastroschisis)
3. Ready to start enteral feeding

Exclusion Criteria:

1. Infants with major congenital anomalies excluding gastrointestinal tract
2. Palliative care patients

4. Septic babies with positive blood, CSF or urine culture

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-12-03 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Intestinal microbiome | 3 weeks after surgury
  Stool microbiome

SECONDARY OUTCOMES:
Length of hospital stay | 6 months
  Time between birth and hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Alixe Howlett, MD, Principal Investigator — University of Calgary; Belal N Alshaikh, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No